CLINICAL TRIAL: NCT05180851
Title: Safety and Efficacy of Recombinant L-IFN Adenovirus Injection in Relapsed/Refractory Solid Tumors: a Single/Multicenter, Dose-increasing, Cohort Extension Clinical Study
Brief Title: Safety and Efficacy of Recombinant Oncolytic Adenovirus L-IFN Injection in Relapsed/Refractory Solid Tumors Clinical Study
Acronym: YSCH-01
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Fengxian District Central Hospital (Other)
Collaborators: Shanghai Yuansong Biotechnology Co., LTD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YSCH-01-0000
Record Dates: First submitted 2021-12-20; First posted 2022-01-06 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Head and Neck Cancer; Melanoma; Breast Cancer; Bladder Cancer; Ovarian Carcinoma; Cervical Carcinoma; Lung Cancer
Keywords: Cancer targetting gene-virotherapy(CTGVT) virus (YSCH-01); Oncolytic virus; Oncolytic adenovirus; Replicative adenovirus
MeSH Terms: conditions — Head and Neck Neoplasms; Melanoma; Breast Neoplasms; Urinary Bladder Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Lung Neoplasms; Virus Diseases | interventions — Oncolytic Virotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safety and efficacy of recombinant L-IFN adenovirus injection in relapsed/refractory solid tumors (Experimental): 1.Only 1 lesion: If the tumor volume is less than or equal to 10 cm3, the whole tumor is injected radially and evenly.
  If the tumor volume was >10 cm3, the tumor was evenly divided into five quadrants and injected into one quadrant at a time.
  2. If there are 2 or more lesions, the most manageable tumor injection is selected; 3. Priority should be given to the body surface metastases that meet the evaluation criteria for tumor efficacy.
  4. According to patients' conditions (e.g., patients with thorax and ascites), the investigator and the research group and cooperative units jointly explored other drug administration approaches (e.g., bladder infusion, thorax and abdominal cavity administration)
  Interventions: Drug: Recombinant L-IFN adenovirus injection

INTERVENTIONS:
Drug: Recombinant L-IFN adenovirus injection — Before use, dilute the product with normal saline according to the size of the tumor to an appropriate volume (10-30% of the total volume of the tumor), or adjust appropriately according to the specific tumor situation, inject directly into the tumor or inject under the guidance of B ultrasound /CT, inject the drug solution into the tumor edge and tumor evenly
  Other Names: (YSCH-01); Cancer targetting gene-virotherapy(CTGVT) virus (YSCH-01); Replicative adenovirus; Oncolytic virus; Oncolytic adenovirus

SUMMARY:
This is an open-label, dose escalation study of the safety and tolerability of Recombinant oncolytic adenovirus L-IFN injection（YSCH-01） when administered via intratumoral injection in patients with advanced solid tumors. The purpose of this study is to assess the safety and tolerability of Recombinant L-IFN adenovirus injectionand to determine the recommended phase 1 dose for further study. The study will also evaluate antitumor activity, objective response rate, pharmacokinetics and virus shedding of Recombinant L-IFN adenovirus injection

DETAILED DESCRIPTION:
This is an investigator initiated , open-label, study of Recombinant oncolytic adenovirus L-IFN injection given via intratumoral (IT) injection as a single agent in participants with advanced solid tumors. The study is a single agent dose escalation which will use a 3+3 design to evaluate escalating doses of Recombinant L-IFN adenovirus injection. Total enrollment will depend on the toxicities and/or activity observed, with approximately19-28 evaluable participants enrolled.

The primary study objective is to determine the safety, tolerability, and maximum tolerated dose (MTD) of intratumoral administration of Recombinant oncolytic adenovirus L-IFN injection as a single agent. Secondary objectives will assess efficacy overall response rate, as well as disease control rate, progression free survival, duration of response, and anti-tumor immune responses.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 and ≤ 75 years;
2. Patients with advanced malignant solid tumors, histologically or cytologically confirmed, who have failed standard therapy, have no standard therapy, are not eligible for standard therapy at this stage, or have refused standard therapy；
3. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1), the length of non-lymph node lesion ≥10 mm or the short diameter of lymph node lesion ≥15 mm according to CT or MRI cross-sectional images;CT scan of the longest axis of measurable lesions ≥10 mm (CT scan thickness ≤5 mm)；
4. There were injectable tumor lesions that met the requirements of the current dose group, including superficial lesions and deep lesions that could be injected under the guidance of B-ultrasound /CT；
5. ECOG score of 0 ~ 2;
6. Sufficient hematopoietic capacity: ANC ≥1.0 ×10^9/L (no short-acting albino within 1 week, no long-acting albino within 2 weeks), platelet count ≥75 ×10^9/L, HGB > 80 g/L (no blood transfusion within 2 weeks)；
7. Adequate liver and kidney function: AST and ALT ≤3 times ULN in patients without liver metastasis, ≤5 times ULN in patients with liver metastasis; Total bilirubin ≤1.5 ULN (excluding hyperbilirubinemia or hyperbilirubin of non-liver origin);Creatinine ≤2.0 ULN and creatinine clearance and creatinine clearance ≥40 mL/min;
8. Eligible and fertile patients (male and female) must agree to use a reliable contraceptive method during the trial and for at least 90 days after the last dose; Women of childbearing age (15-49 years) must have a negative pregnancy test within 7 days before starting treatment;
9. PT or INR <1.5 ULN, and APTT <1.5 ULN；
10. Expect to live at least 12 weeks；

Exclusion Criteria:

1. Received any antineoplastic therapy within 2 weeks prior to initial treatment；
2. Systemic diseases that have not been stably controlled after treatment, such as diabetes, serious organic cardiovascular and cerebrovascular diseases, cardiac insufficiency, hypertension, heart block above ⅱ degree, myocardial infarction within 6 months, cerebral infarction within 6 months, etc.
3. Pregnancy or lactation;
4. Uncontrolled infectious diseases, such as baseline HBV DNA≥2000 IU/ml, anti-HIV positive, HCV-RNA positive;
5. Other active infections of significant clinical significance;
6. Subjects with other active malignancies within the past 5 years, such as basal or squamous skin cancer, superficial bladder cancer, or breast cancer in situ, that have been completely cured and do not require follow-up treatment are excluded;
7. Severe autoimmune diseases such as ulcerative colitis, Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus, autoimmune vasculitis, or Wegener's granuloma require long-term (more than 2 months) systemic immunosuppressive therapy, but subjects with the following conditions are admitted:

   Autoimmune hypothyroidism requiring only hormone replacement therapy; Skin disorders that do not require systemic treatment (e.g., eczema, a rash of less than 10% of the body surface);
8. Subjects with allergic constitution, allergy to immunotherapy or related drugs;
9. Organ failure; Coronary heart: grades ⅲ and ⅳ;Or hypertension that cannot be controlled by standard treatment, a history of myocarditis or myocardial infarction within one year; Gallo liver: achieves grade C on the Child-Turcotte-Pugh liver function scale; Gallonic kidney: renal failure and uremia; Lung: symptoms of severe respiratory failure; Brain unconsciously: people with consciousness disorder have active brain metastases;
10. Patients with active bleeding and thrombotic diseases requiring treatment;
11. Patients with uncontrollable pleural and abdominal effusion requiring clinical treatment or intervention;
12. Subjects requiring systemic corticosteroids (equivalent to >10 mg prednisone/day) within 14 days prior to enrollment or during the study period;

    The following conditions are allowed to join the group:

    Allow subjects to use topical or inhaled corticosteroids; Allows short-term (≤7 days) use of glucocorticoids for the prevention or treatment of non-autoimmune allergic diseases;
13. Subject suffering from any mental illness, including dementia, altered mental state, that may affect informed consent and understanding of the relevant questionnaire;
14. Participated in clinical trials of other drugs or medical devices within 4 weeks;
15. If the investigator determines that they have a serious and uncontrollable disease or other conditions that may affect their acceptance of this study, they are not considered suitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Up to 28 days
  To define the maximum tolerated dose (MTD) of intratumoral administration of Recombinant L-IFN adenovirus injection in humans with malignant tumors.
Safety and tolerability assessed by Adverse Events (AEs) | Time Frame: Up to 6 months
  An AE is any untoward medical occurrence in a subject administered an investigational product (IP), and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP whether or not considered related to the IP

SECONDARY OUTCOMES:
Number of participants with vital sign abnormalities and /or adverse event | Up to 6 months
  Number of participants with potentially clinically significant laboratory values
Number of participants with laboratory value abnormalities and/or adverse events | Up to 6 months
  Number of participants with potentially clinically significant laboratory values
Presence of neutralizing antibodies of antidrug antibodies (ADAs) development | Up to 6 months
  To evaluate the immunogenicity of Recombinant L-IFN adenovirus injection given as single agent post injection

CONTACTS AND LOCATIONS:
Overall Officials: Rong Zhang, MD, Principal Investigator — Shanghai Fengxian District Central Hospital
Locations (1):
- Shanghai Fengxian District Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] He Y, Huang X, Li X, Liu H, Liu M, Tao J, Shan Y, Raza HK, Liu Y, Zhong W, Cao XP, Yang YY, Li R, Fang XL, Zhang KJ, Zhang R, Liu F. Preliminary efficacy and safety of YSCH-01 in patients with advanced solid tumors: an investigator-initiated trial. J Immunother Cancer. 2024 May 7;12(5):e008999. doi: 10.1136/jitc-2024-008999. PMID 38719544